CLINICAL TRIAL: NCT05116501
Title: Novel Insights Into the Genetic Background of Patients With Low Von Willebrand Factor Levels Using Next-generation Sequencing
Brief Title: Genetic Background of Patients With Low Von Willebrand Factor Levels
Acronym: LOVMIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2392
Record Dates: First submitted 2021-09-27; First posted 2021-11-11 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2021-09

CONDITIONS: Low Von Willebrand Factor
Keywords: von Willebrand factor; VWF; Von Willebrand disease; VWD; Low VWF; NGS; Whole exome sequencing
MeSH Terms: conditions — von Willebrand Diseases | interventions — Exome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low VWF (Experimental): In patients with low VWF levels, whole-exome sequencing will be performed to identity possible variants in the VWF gene or other genes that are associated with reduced VWF plasma levels. Furthermore, a correlation study between variants identified and the bleeding symptoms of patients will be performed.
  Interventions: Diagnostic Test: Whole-exome sequencing
- Healthy controls (Other): In healthy controls, the investigators will analyze the whole-exome sequencing to include the variants that are either not present in healthy controls or are present but with a significantly lower frequency than the patients.
  Interventions: Diagnostic Test: Whole-exome sequencing

INTERVENTIONS:
Diagnostic Test: Whole-exome sequencing — Whole Exome Sequencing (WES), as a comprehensive genetic test, will be used to identify changes in a patient's DNA that are causative or related to patient's low VWF levels.

SUMMARY:
Von Willebrand disease (VWD) is caused by either quantitative or qualitative von Willebrand (VWF) defects and is the commonest inherited bleeding disorder with an estimated prevalence of about 1% in the general population. According to several guidelines, patients with a mild quantitative reduction in VWF (30-50 IU/dL) should be labeled as "low VWF". Quantitatively VWF defects account for almost 75% of all cases with VWD and among them, low VWF seems to be the most common form. Studies on patients with VWD reported only around 50% VWF mutations in low VWF cases indicating that some possible genes outside of the VWF gene may be responsible for the low VWF levels. To date, using genome-wide association study (GWAS) more than 19 non-VWF loci (such as ABO blood group system, Stabilin 2, Scavenger Receptor Class A Member 5, C-Type Lectin Domain Family 4 Member M, etc.) were identified to be associated with VWF levels. The identified genes are related to different mechanisms of the VWF life-cycle such as synthesis, secretion, glycosylation, or clearance. Despite the importance of the genetic background of low VWF levels for understanding its etiology, this issue is not well investigated yet. Thus the Low VWF Milan Cohort (LOVMIC) Study is designed to address some unanswered questions in patients with low VWF.

DETAILED DESCRIPTION:
Despite the absence of mutation in the VWF gene in a significant number of individuals with reduced VWF levels and also the lack of knowledge for the responsible mechanisms, this study sought to determine the following goals:

* Evaluation of the genetic background of low VWF level dilemma and identifying the gene (s) outside of the VWF gene that is associated with decreased VWF levels.
* Evaluating the correlation between candidate variants and patients' bleeding manifestations.

Study design:

Non-pharmacological Interventional National Monocentric Study. Promoter: Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico Coordinating center and patient recruitment unit: Department of General Medicine - Hemostasis and Thrombosis - Angelo Bianchi Bonomi Hemophilia and Thrombosis Center

Setting: outpatients' clinic

The study population will be selected from the referral adult patients/healthy controls to the A. Bianchi Bonomi Hemophilia and Thrombosis Center in Fondazione IRCCS Ca' Granda Maggiore Policlinic hospital.

Recruiting method:

Selected patients (base on the previous laboratory results) will be invited to participate in the study by physicians at the center through phone calls. Also, normal controls (age- and sex-matched with patients) will be enrolled in the study. Data regarding the healthy controls will be obtained either from the available public database or obtained by evaluation of collected samples from the normal subjects who have been selected by the A. Bianchi Bonomi Hemophilia and Thrombosis Center.

Enrolment, visit, and blood samples collection:

Following the agreement of patients for participating in the study and signing the informed consent, 3 tubes (each 3.5 ml) of the blood sample will be collected for performing VWD-related laboratory tests (VWF antigen (VWF:Ag), VWF ristocetin cofactor (VWF:RCo), Factor VIII clotting assay (FVIII:C)) and Whole-exome sequencing (WES). In addition, a routinely clinical examination will be done by specialized physicians, according to a Case Report Form (CRF) to collect the data regarding age, sex, blood group, and clinical manifestations including the International Society on Thrombosis and Haemostasis Bleeding Assessment Tool (ISTH-BAT).

Genetic analysis:

* Genomic DNA will be extracted using the automated instrument from QIAGEN available in the central genetic laboratory at the Fondazione IRCCS Ca' Granda Maggiore Policlinic hospital
* WES will be performed on all samples using NextSeq 2000 instrument in the central genetic laboratory at the Fondazione IRCCS Ca' Granda Maggiore Policlinic hospital.
* Data will be analyzed following the same strategy in both cases and controls. First, the VWF gene will be evaluated. Then, the analysis will be extended to the other genes that were previously described as related to VWF level variations. Lastly, exome data will be considered.
* The association between VWF levels and candidate variants will be assessed.
* All analyses will be performed considering variants' minor allele frequency (MAF), age, sex, ABO to control for confounding.

ELIGIBILITY:
Inclusion Criteria for patients:

* Adult patients who were diagnosed with "low VWF" and have VWF:Ag and/or VWF:RCo between 30-50 IU/dL with a ratio of VWF:RCo/VWF:Ag > 0.6.
* Subjects who have given informed consent to participate in the study according to the Declaration of Helsinki

Inclusion Criteria for healthy controls:

* Healthy subjects with no known bleeding disorders and with negative thrombophilia screening results
* Subjects who have given informed consent to participate in the study according to the Declaration of Helsinki

Exclusion Criteria:

* Pregnant women
* Patients with acquired von Willebrand disease syndrome

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Genetic variants in the VWF gene or other genes associated with low VWF plasma levels | 8 months after starting the project
  More than 19 different genes have been identified by genome-wide association studies that affect the plasma VWF levels. These genes (in addition to VWF) are including STXBP5, SCARA5, ABO, STAB2, STX2, TCN2, CLEC4M, PDHB/PXK/KCTD6, SLC39A8, FCHO2/TMEM171/TNPO1, HLA, GIMAP7/GIMAP4, OR13C5/NIPSNAP, DAB2IP, C2CD4B, RAB5C-KAT2A, TAB1/SYNGR1, and ARSA. Some studies showed an association between specific variants with a minor allele frequency (MAF) > 10% and the reduction of VWF levels or severe clinical symptoms in patients with VWD.
  As a primary outcome, whole-exome sequencing will be carried out in 300 subjects (150 patients and 150 healthy controls) to identify variants either in the VWF gene or the aforementioned genes or some new genes that are associated with reduced VWF levels in plasma.

SECONDARY OUTCOMES:
Correlation between the bleeding presentation and identified variants in patients with low VWF | 12 months after starting the project
  As the second outcome, the association between the identified potential variants and patient bleeding manifestations will be evaluated. The ISTH-BAT is used to quantify bleeding symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Flora Peyvandi, MD, PhD, Principal Investigator — A.Bonomi Hemophilia and Thrombosis Center, Foundation IRCCS Ca' Granda Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, A.B.Bonomi Hemophilia and Thrombosis Center, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
All data, including exposure and outcomes, will be collected based on a Case report form (CRF) and thereafter they will be reported on a computer database. Each process to promote data quality will be guaranteed. In particular, data insertion and correction will be performed by the principal investigator (PI) or by those investigators designated by the PI and all data will be securely stored to ensure complete pseudonymization. The insertion of all the data in the CRF and the computer database will be performed correctly and accurately according to the source documentation (medical reports and records). In case of a lack of data, and accurate motivation will be provided (not available/not requested from the patient).

REFERENCES:
- [Background] James PD, Connell NT, Ameer B, Di Paola J, Eikenboom J, Giraud N, Haberichter S, Jacobs-Pratt V, Konkle B, McLintock C, McRae S, R Montgomery R, O'Donnell JS, Scappe N, Sidonio R, Flood VH, Husainat N, Kalot MA, Mustafa RA. ASH ISTH NHF WFH 2021 guidelines on the diagnosis of von Willebrand disease. Blood Adv. 2021 Jan 12;5(1):280-300. doi: 10.1182/bloodadvances.2020003265. PMID 33570651
- [Result] Rodeghiero F, Castaman G, Dini E. Epidemiological investigation of the prevalence of von Willebrand's disease. Blood. 1987 Feb;69(2):454-9. PMID 3492222
- [Result] Laffan MA, Lester W, O'Donnell JS, Will A, Tait RC, Goodeve A, Millar CM, Keeling DM. The diagnosis and management of von Willebrand disease: a United Kingdom Haemophilia Centre Doctors Organization guideline approved by the British Committee for Standards in Haematology. Br J Haematol. 2014 Nov;167(4):453-65. doi: 10.1111/bjh.13064. Epub 2014 Aug 12. No abstract available. PMID 25113304
- [Result] Lavin M, Aguila S, Schneppenheim S, Dalton N, Jones KL, O'Sullivan JM, O'Connell NM, Ryan K, White B, Byrne M, Rafferty M, Doyle MM, Nolan M, Preston RJS, Budde U, James P, Di Paola J, O'Donnell JS. Novel insights into the clinical phenotype and pathophysiology underlying low VWF levels. Blood. 2017 Nov 23;130(21):2344-2353. doi: 10.1182/blood-2017-05-786699. Epub 2017 Sep 15. PMID 28916584
- [Result] Flood VH, Christopherson PA, Gill JC, Friedman KD, Haberichter SL, Bellissimo DB, Udani RA, Dasgupta M, Hoffmann RG, Ragni MV, Shapiro AD, Lusher JM, Lentz SR, Abshire TC, Leissinger C, Hoots WK, Manco-Johnson MJ, Gruppo RA, Boggio LN, Montgomery KT, Goodeve AC, James PD, Lillicrap D, Peake IR, Montgomery RR. Clinical and laboratory variability in a cohort of patients diagnosed with type 1 VWD in the United States. Blood. 2016 May 19;127(20):2481-8. doi: 10.1182/blood-2015-10-673681. Epub 2016 Feb 9. PMID 26862110
- [Result] Sabater-Lleal M, Huffman JE, de Vries PS, Marten J, Mastrangelo MA, Song C, Pankratz N, Ward-Caviness CK, Yanek LR, Trompet S, Delgado GE, Guo X, Bartz TM, Martinez-Perez A, Germain M, de Haan HG, Ozel AB, Polasek O, Smith AV, Eicher JD, Reiner AP, Tang W, Davies NM, Stott DJ, Rotter JI, Tofler GH, Boerwinkle E, de Maat MPM, Kleber ME, Welsh P, Brody JA, Chen MH, Vaidya D, Soria JM, Suchon P, van Hylckama Vlieg A, Desch KC, Kolcic I, Joshi PK, Launer LJ, Harris TB, Campbell H, Rudan I, Becker DM, Li JZ, Rivadeneira F, Uitterlinden AG, Hofman A, Franco OH, Cushman M, Psaty BM, Morange PE, McKnight B, Chong MR, Fernandez-Cadenas I, Rosand J, Lindgren A; INVENT Consortium; MEGASTROKE Consortium of the International Stroke Genetics Consortium (ISGC); Gudnason V, Wilson JF, Hayward C, Ginsburg D, Fornage M, Rosendaal FR, Souto JC, Becker LC, Jenny NS, Marz W, Jukema JW, Dehghan A, Tregouet DA, Morrison AC, Johnson AD, O'Donnell CJ, Strachan DP, Lowenstein CJ, Smith NL. Genome-Wide Association Transethnic Meta-Analyses Identifies Novel Associations Regulating Coagulation Factor VIII and von Willebrand Factor Plasma Levels. Circulation. 2019 Jan 29;139(5):620-635. doi: 10.1161/CIRCULATIONAHA.118.034532. PMID 30586737